CLINICAL TRIAL: NCT06830200
Title: Clinical and Immunological Evaluation of the Efficacy of Chitosan Brush in Non-Surgical Peri-implantitis Treatment
Brief Title: Peri-implantitis Treatment With Chitosan Brush
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Buket Acar, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-23071
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Peri-implantitis
Keywords: Chitosan Brush; Non-Surgical Peri-implantitis Treatment; Peri-implantitis; Cytokine; Titanium Curette
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chitosan Brush (Active Comparator): The implants in the chitosan brush group will be debrided with a chitosan brush dipped in sterile physiological saline solution using a rotary instrument system for 2 minutes. After mechanical treatment, the peri-implant pockets will be washed with sterile physiological saline solution. In cases with BOP+ and PD≥ 4 mm at 3 and 6 months after treatment, the treatment will be repeated in the same way as the previous one. Local infiltration anesthesia will be applied to the patients when deemed necessary. The prosthetic superstructures of the implants will not be removed for clinical examination or treatment. In cases where there is more than one implant in the same patient requiring peri-implantitis treatment, all of these implants will be included in the same treatment group.
  Interventions: Procedure: Non-surgical periodontal treatment with chitosan brush
- Titanium Curette (Active Comparator): The implants in the titanium curette group will be treated with titanium curettes for 2 minutes. After mechanical treatment, the peri-implant pockets will be washed with sterile physiological serum. In cases with BOP+ and PD≥ 4 mm at 3 and 6 months after treatment, the treatment will be repeated in the same way as the previous one. Local infiltration anesthesia will be applied to the patients when deemed necessary. The prosthetic superstructures of the implants will not be removed for clinical examination or treatment. In cases where there is more than one implant requiring peri-implantitis treatment in the same patient, all of these implants will be included in the same treatment group.
  Interventions: Device: Non-surgical treatment of pre-implantitis with titanium curette

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment with chitosan brush — Non-surgical treatment of pre-implantitis with chitosan brush
  Arms: Chitosan Brush
Device: Non-surgical treatment of pre-implantitis with titanium curette — Description: Non-surgical treatment of pre-implantitis with titanium curette
  Arms: Titanium Curette

SUMMARY:
In dentistry, dental implant applications for tooth loss/deficiency are prominent and provide successful long-term results in terms of functionality and aesthetics. However, peri-implant diseases such as peri-implant mucositis and peri-implantitis may develop due to biofilm accumulation around the implant. In peri-implantitis, in addition to the clinical inflammation findings seen in peri-implant mucositis, there is also progressive bone loss. This condition is to be treated with non-surgical or surgical methods. Titanium curettes, ultrasonic instruments, laser systems, and chitosan brushes are used for biofilm removal in non-surgical treatment. Chitosan is a natural polysaccharide obtained from chitin. It is biocompatible, biodegradable, and has antibacterial activity. In addition, chitosan reduces the levels of IL-1β, IL-6, and TNF-α, which also play a role in the pathogenesis of peri-implantitis, and exhibits anti-inflammatory effects on macrophages activated by lipopolysaccharide. Although many methods are used to treat peri-implantitis, successful and predictable results cannot be obtained. This study aims to examine the clinical and immunological findings and observe the changes in the non-surgical treatment of peri-implantitis using chitosan brush or titanium curette over 12 months. Sixty dental implants diagnosed with peri-implantitis clinically and radiographically at the Department of Periodontics, Faculty of Dentistry, Hacettepe University will be included in the study. Non-surgical peri-implantitis treatment of these patients will be performed using a chitosan brush (N=30, case group) or titanium curette (N=30, control group). Pre-operative and post-operative 3rd, 6th, and 12th months, clinical periodontal indices will be recorded, peri-implant crevicular fluid (PIF) will be collected, and maintenance treatment will be applied to the patients. IL-1β, TNF-α, IL-8, IL-10, and IL-17 levels in the collected PIF will be determined by the ELISA method. The effectiveness of chitosan brush and titanium curette in treating peri-implantitis will be evaluated and compared clinically and immunologically.

ELIGIBILITY:
Inclusion Criteria:

* Presence of peri-implantitis in an implant that has been in function for more than 12 months
* Age ≥ 18 and < 65
* Agreeing to participate in the study after reading the informed consent form
* Completion of periodontal treatment of patients diagnosed with periodontitis before inclusion in the study

Exclusion Criteria:

* Patients under 18 years of age
* Patients who have received or are currently receiving radiotherapy, chemotherapy and long-term systemic corticosteroid treatment
* Patients who received systemic antibiotics within 6 months from baseline
* Pregnant or lactating patients
* Patients with anatomical abnormalities around the implant (e.g., apically positioned implants adjacent to a tooth)
* Patients with prostheses that prevent access for implant debridement with chitosan brushes or titanium curettes
* Implants with an overdenture superstructure
* Implants to be explanted
* Patients with ASA score ≥ 3
* Patients reporting reactions or adverse events to chitosan, stainless steel, adhesives, or polypropylene
* Clinically mobile implants
* Recently placed and non-osseointegrated implants
* Around major nerves and blood vessels, if there is a risk of structural damage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Probing Pocket Depth | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  The distance between the mucosal margin and the bottom of the peri-implant pocket [six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual and distolingual) on each implant]
Radiographic Bone Level (RBL) | From the baseline to the 12th month (Baseline, 6th, 12th months)
  RBL is determined in millimeters by metrically measuring the distance from the implant shoulder to the first bone-implant contact on the radiograph. Increasing RBL indicates worse outcome

SECONDARY OUTCOMES:
Gingival index (GI) | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  According to the GI system; 0: Normal gingiva
  1. Mild inflammation with no edema, color change or bleeding on probing in the gingiva
  2. Moderate inflammation with redness, edema and brightness in the gingiva and bleeding on probing
  3. Severe inflammation with significant redness, edema, ulceration and spontaneous bleeding.
  Six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual and distolingual) on each implant. The gingival index of an implant is calculated by dividing the total score of that implant by 4. Increased GI indicates worse outcome.
Plaque Index (PI) | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  According to PI scores; 0: No plaque
  1. Invisible film-like plaque attached to the free gingival margin and adjacent implant surface, detectable with a probe
  2. Visible, moderate soft attachment within the gingival pocket or on the gingival margin and adjacent implant surface
  3. Indicates the presence of dense soft attachment within the gingival pocket or on the gingival margin and adjacent implant surface.
  Six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual and distolingual) were measured on each implant.The arithmetic average of 4 measurement values obtained from an implant is recorded as the PI score for that implant. Increased PI indicates worse outcome
Bleeding on Probing | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
Keratinized Mukoza Width | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  The distance between the keratinized mucosa margin and the mucogingival junction in the mid-buccal region of the implant
Recession Depth | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  The distance between the margin of the prosthetic restoration and the keratinized mucosal marjin
IL-1β | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  From PIOS
TNF-α | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  From PIOS
IL-8 | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  From PIOS
IL-10 | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  From-PIOS
IL-17 | From the baseline to the 12th month (Baseline, 3rd, 6th, 12th months)
  From PIOS

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)